CLINICAL TRIAL: NCT05997303
Title: Continuous Norepinephrine Administration and Blood Pressure Stability During Anesthetic Induction - A Randomized Controlled Trial
Brief Title: Continuous Norepinephrine Administration and Blood Pressure Stability During Anesthetic Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-101053-BO-ff
Record Dates: First submitted 2023-07-17; First posted 2023-08-18 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Blood Pressure; Perioperative Hypotension
Keywords: blood pressure stability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous norepinephrine administration (Other): continuous norepinephrine infusion via an infusion pump; norepinephrine dose will be at the discretion of the treating anesthesiologists
  Interventions: Other: Continuous norepinephrine infusion via an infusion pump
- Manual bolus norepinephrine administration (Other): manual bolus norepinephrine administration; norepinephrine dose will be at the discretion of the treating anesthesiologists
  Interventions: Other: Manual bolus norepinephrine administration

INTERVENTIONS:
Other: Continuous norepinephrine infusion via an infusion pump — Patients will be randomized 1:1 to continuous norepinephrine infusion via an infusion pump or to manual bolus norepinephrine administration. The norepinephrine dose will be at the discretion of the treating anesthesiologists.
  Arms: Continuous norepinephrine administration
Other: Manual bolus norepinephrine administration — Patients will be randomized 1:1 to continuous norepinephrine infusion via an infusion pump or to manual bolus norepinephrine administration. The norepinephrine dose will be at the discretion of the treating anesthesiologists.
  Arms: Manual bolus norepinephrine administration

SUMMARY:
This is a randomized trial investigating whether continuous norepinephrine administration via an infusion pump - compared to manual bolus administration - increases blood pressure stability within the first 15 minutes of anesthetic induction in non-cardiac surgery patients.

The secondary endpoints area under a MAP of 65, 60, 50, and 40 mmHg [mmHg × min], cumulative duration of a MAP <65, <60, <50, and <40 mmHg [min], area above a MAP of 100, 110, 120, and 140 mmHg [mmHg min], cumulative duration of a MAP >100, >110, >120, and >140 mmHg [min] and cumulative dose of norepinephrine indexed to body weight [μg/kg] within the first 15 minutes of anesthetic induction will be assessed.

DETAILED DESCRIPTION:
not provided

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 45 years
* American Society of Anesthesiologists physical status II-IV
* scheduled for elective major non-cardiac surgery under general anesthesia
* continuous intraarterial blood pressure monitoring using a radial arterial catheter for clinical indications not related to the trial
* sinus rhythm

Exclusion Criteria:

* Clinical indication to use a continuous norepinephrine infusion via an infusion pump during anesthetic induction
* Need for femoral artery catheterization
* History of intracranial bleedings or aneurysms
* Patients who are incapable of giving consent
* Pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Blood pressure stability | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  Generalized average real variability (gARV) of mean arterial pressure (MAP) within the first 15 minutes of anesthetic induction [mmHg/min]; the gARV is the sum of absolute values of the differences between neighboring measurements for all measurements divided by the total measurement duration in [mmHg/min].

SECONDARY OUTCOMES:
Area under MAP | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  Area under a MAP of 65, 60, 50, and 40 mmHg [mmHg × min]. MAP will be measured using intraarterial blood pressure monitoring.
Cumulative duration of a MAP below | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  Cumulative duration of a MAP <65, <60, <50, and <40 mmHg [min]. MAP will be measured using intraarterial blood pressure monitoring.
Area above MAP | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  Area above a MAP of 100, 110, 120, and 140 mmHg [mmHg × min]. MAP will be measured using intraarterial blood pressure monitoring.
Cumulative duration of a MAP above | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  Cumulative duration of a MAP >100, >110, >120, and >140 mmHg [min]. MAP will be measured using intraarterial blood pressure monitoring.
Cumulative dose of norepinephrine | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  Cumulative dose of norepinephrine indexed to body weight [μg/kg]

OTHER OUTCOMES:
Explorative aim - effect on (advanced) hemodynamic variables - stroke volume index | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  We aim to investigate the effect of giving norepinephrine continuously via an infusion pump during anesthetic induction on stroke volume index [ml/m^2] using invasive uncalibrated pulse wave analysis (MostcareUP System).
Explorative aim - effect on (advanced) hemodynamic variables - heart rate | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  We aim to investigate the effect of giving norepinephrine continuously via an infusion pump during anesthetic induction on heart rate [beats/minute] using invasive uncalibrated pulse wave analysis (MostcareUP System).
Explorative aim - effect on (advanced) hemodynamic variables - cardiac index | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  We aim to investigate the effect of giving norepinephrine continuously via an infusion pump during anesthetic induction on cardiac index [l/min/m^2] using invasive uncalibrated pulse wave analysis (MostcareUP System).
Explorative aim - effect on (advanced) hemodynamic variables - systemic vascular resistance index | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  We aim to investigate the effect of giving norepinephrine continuously via an infusion pump during anesthetic induction on systemic vascular resistance index [dyn × s × cm^-5 × m^2] using invasive uncalibrated pulse wave analysis (MostcareUP System).
Explorative aim - effect on (advanced) hemodynamic variables - pulse pressure variation | Measurement period of 15 minutes starting at the beginning of the anesthetic induction
  We aim to investigate the effect of giving norepinephrine continuously via an infusion pump during anesthetic induction on pulse pressure variation [%] using invasive uncalibrated pulse wave analysis (MostcareUP System).

CONTACTS AND LOCATIONS:
Overall Officials: Christina Vokuhl, M.D., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vokuhl C, Kouz K, Flick M, Krause L, Kroker A, Moll-Khosrawi P, Zollner C, Sessler DI, Saugel B, Thomsen KK. Continuous versus bolus norepinephrine administration and arterial blood pressure stability during induction of general anaesthesia in high-risk noncardiac surgery patients: a randomised trial. Br J Anaesth. 2025 Oct;135(4):878-885. doi: 10.1016/j.bja.2025.06.025. Epub 2025 Jul 30. PMID 40744797